CLINICAL TRIAL: NCT05756062
Title: Antioxidant and Anti-inflammatory Effects of Oral Supplementation With a Highly-Concentrated Docosahexaenoic Acid (DHA) Triglyceride in Patients With Keratoconus: A Randomized Controlled Preliminary Study
Brief Title: Supplementation With a Highly-Concentrated Docosahexaenoic Acid (DHA) Triglyceride in Patients With Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Cristina Peris, Head Unit of Cornea and Anterior Eye Diseases, FISABIO Medical Ophthalmology (FOM), Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI_77
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA group (Experimental): Supplementation with a highly-concentrated docosahexaenoic acid (DHA) triglyceride (1000 g/day) for 3 months
  Interventions: Dietary Supplement: Highly-concentrated DHA triglyceride (Tridocosahexanoin-AOX 70%)
- Control group (No Intervention): Routine care

INTERVENTIONS:
Dietary Supplement: Highly-concentrated DHA triglyceride (Tridocosahexanoin-AOX 70%) — Daily administration of 2 capsules of the study product (1000 mg DHA triglyceride) for 3 months
  Arms: DHA group

SUMMARY:
The goal of this randomized controlled preliminary study is to assess the effect of daily supplementation with a nutraceutical formulation of a highly-concentrated DHA triglyceride plus minerals on ophthalmological parameters and biomarkers of oxidative stress and inflammation in blood samples of patients with keratoconus.The main questions it aims to answer are:

* Improvements in ophthalmological parameters.
* Increase in antioxidant capacity, decrease in inflammatory status, and changes in lipidomic biomarkers.

Participants are patients with keratoconus who will be given the nutraceutical supplementation for 3 months.

If there is a comparison group: Researchers will compare patients with keratoconus not given the nutraceutical formulation to see differences in the study variables

DETAILED DESCRIPTION:
Among omega-3 polyunsaturated fatty acids (PUFAs), docosahexaenoic acid (DHA, C22:6-n3), a critical component of cell membrane phospholipids, exerts pleiotropic effects at both central and peripheral levels with health benefits in many aspects of neuronal, immune, cognitive, and cardiovascular functions Clinical studies of dietary sup-plementation with a highly-concentrated DHA triglyceride have shown consistent an-ti-inflammatory, antioxidant, antiangiogenic, and antiproliferative effects targeting pathophysiological pathways involved in different eye diseases, including diabetic retinopathy and macular edema, ocular surface disorders, meibomian gland dysfuncton, and pseudoexfoliative glaucoma.

Based on this experience, it was considered of interest to explore the antioxidant and anti-inflammatory potential of a highly-concentrated DHA triglyceride supplement in patients with keratoconus. For this purpose, a prospective preliminary study was designed to assess the effects of 3-month DHA nutritional supplementation on clinical variables, and inflammatory and oxidative stress biomarkers of patients with early and moderate keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus stages I to III according to the Amsler-Krumeich classification
* Non-contact lens wearers
* No history of previous corneal surgery
* Capacity to volunteer and willing and able to follow the study protocol

Exclusion Criteria:

* Advanced keratoconus (stage IV of the Amsler-Krumeich classification
* Other ectasias (e.g. iatrogenic secondary to ocular surface surgery with excimer laser, radial keratotomy, traumatic corneal ectasia, etc.)
* Eyelid alterations
* Previous ocular surgery
* Any ocular or systemic condition that may affect the interpretation of results
* Glaucoma or ocular hypertension
* History of ocular trauma, infection or inflammation
* Current treatment with topical or anti-inflammatory drugs
* Use of nutritional supplements including omega-3 fatty acids, vitamins and minerals (unless a washout period of 1 month had been established)
* Hypersensitivity to fish proteins
* Pregnant women
* Refusal to sign the written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Corneal topography | Baseline and after 3 months of supplementation (end of study)
  Changes of ophthalmological parameters
Antioxidant variables | Baseline and after 3 months of supplementation (end of study)
  Changes in plasma total antioxidant capacity (TAC), malondialdehyde (MDA) and glutathione (GSH), and GSH/GSSH ratio
Anti-inflammatory variables | Baseline and after 3 months of supplementation (end of study)
  cytokine levels IL-1beta, IL-4, IL-6, IL-10, IL-18, TNFalpha, VEGF-A

SECONDARY OUTCOMES:
Lipidomic variables | Baseline and after 3 months of supplementation (end of study)
  Serum levels of DHA, arachidonic acid (ARA), n-6 PUFA/n-3 PUFA, omega-3 index

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Peris-Martinez, MD, Principal Investigator — FISABIO Medical Ophthalmology (FOM)
Locations (1):
- FISABIO Medical Ophthalmology (FOM), Valencia, Spain

IPD SHARING:
Plan to Share IPD: No